CLINICAL TRIAL: NCT00207675
Title: A Randomized, Multicenter, Open-label Study to Evaluate the Safety and Efficacy of Anti-TNF a Chimeric Monoclonal Antibody (Infliximab, REMICADE) in Pediatric Subjects With Moderate to Severe CROHN'S Disease.
Brief Title: A Study of the Safety and Efficacy of Infliximab (Remicade) in Pediatric Patients With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Centocor BV (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CR004786
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-03

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; pediatric Crohn's Disease
MeSH Terms: conditions — Crohn Disease; Pediatric Crohn's disease | interventions — Infliximab

INTERVENTIONS:
Drug: infliximab

SUMMARY:
A study of the safety and efficacy of infliximab (Remicade) in pediatric patients with moderate to severe Crohn's Disease

DETAILED DESCRIPTION:
This is a medical research study to evaluate the safety and effectiveness of an antibody called infliximab (Remicade) in the treatment of children with Crohn's disease. In this study, subjects will receive multiple doses of infliximab over 62 weeks. The goal of the study is to ensure that the medication is safe and effective in children when it is given for an extended period of time. All subjects will receive an induction regimen of 5 mg/kg infliximab at Weeks 0, 2, and 6. Subjects will then receive either 5 or 10 mg/kg infliximab either every 8 or 12 weeks for up to 46 weeks followed by an open label extension for up to three additional years.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 6 and 17 years
* Have had Crohn's disease diagnosed for at least 3 months prior to screening, with gastritis, duodenitis, colitis, ileitis, or ileocolitis, previously confirmed by endoscopy and biopsy
* Have active Crohn's disease despite adequate current treatment with an immunomodulator (ie, AZA, 6-MP, or MTX).

Exclusion Criteria:

* Disease complications for which surgery might be indicated
* Surgery for bowel diversion with placement of a stoma within 3 months prior to screening
* Positive stool examination for enteric pathogens including Giardia lamblia, Clostridium difficile, Shigella species, and Salmonella species.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2003-02; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Clinical response at Week 10, defined as a decrease from baseline in the PCDAI score of at least 15 points with a total score of no more than 30 points at Week 10.

SECONDARY OUTCOMES:
Clinical response at Week 54; Clinical remission at Week 54; Change from baseline in corticosteroid use at Week 54; Change from baseline in height status at Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Hyams J, Crandall W, Kugathasan S, Griffiths A, Olson A, Johanns J, Liu G, Travers S, Heuschkel R, Markowitz J, Cohen S, Winter H, Veereman-Wauters G, Ferry G, Baldassano R; REACH Study Group. Induction and maintenance infliximab therapy for the treatment of moderate-to-severe Crohn's disease in children. Gastroenterology. 2007 Mar;132(3):863-73; quiz 1165-6. doi: 10.1053/j.gastro.2006.12.003. Epub 2006 Dec 3. PMID 17324398
- [Result] Thayu M, Leonard MB, Hyams JS, Crandall WV, Kugathasan S, Otley AR, Olson A, Johanns J, Marano CW, Heuschkel RB, Veereman-Wauters G, Griffiths AM, Baldassano RN; Reach Study Group. Improvement in biomarkers of bone formation during infliximab therapy in pediatric Crohn's disease: results of the REACH study. Clin Gastroenterol Hepatol. 2008 Dec;6(12):1378-84. doi: 10.1016/j.cgh.2008.07.010. PMID 19081527
- See also: A Randomized, Multicenter, Open-label Study to Evaluate the Safety and Efficacy of Anti-TNFa Chimeric Monoclonal Antibody (Infliximab, REMICADE�) in Pediatric Subjects with Moderate to Severe Crohn's Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=152&filename=CR004786_CSR.pdf
- See also: |A Randomized, Multicenter, Open-label Study to Evaluate the Safety and Efficacy of Anti-TNFa Chimeric Monoclonal Antibody (Infliximab, REMICADE®) in Pediatric Subjects with Moderate to Severe Crohn's Diseas — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=152&filename=CR004786_REF1.pdf